CLINICAL TRIAL: NCT05258227
Title: A Randomized Control Trial To Comapre The Effects Of Proprioceptive Training And Core Instability Strength Training On Balance,Pain And Physical Functions In Patients With Knee Osteoarthritis
Brief Title: Comapre Effects Of Proprioceptive Training And Core Instability Strength Training In Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-FSD-00278
Record Dates: First submitted 2022-02-20; First posted 2022-02-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
Keywords: Proprioceptive Training; Core Instability; Strength Training; Knee Osteoarthritis; Randomized Control Trial; Balance; Physical Functions
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be double blinded as the assessors and the subjects of the study are kept blind towards the treatment group to which patients are allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Strength Training (Experimental): * Conservation physical therapy includes TENS 15 min + Infrared 15 min simultaneously.
  * Proprioceptive strength training for 30 min includes following exercises:
  Strengthening of Quadriceps Ankle extensors and Hip abductors strengthening Zigzag walking Heel to toe walk forward and backwards toe to heel Standing on one leg while holding wall, eyes open and eyes closed
  Interventions: Other: Conservational Physical Therapy and Proprioceptive Strength Training
- Core Instability Strength Training (Experimental): * Conservational therapy includes TENS for 15 min+ Infrared for 15 min simultaneously.
  * Core instability strength training for 30 minutes includes following exercises:
  Quadriceps stretch, crook lying, abdominal hallowing Dynamic Hamstrings stretch Bridging arms at side Crook lying+lifting both legs at right angle with hands resting on thighs
  Interventions: Other: Conservational Physical Therapy and Core Instability Strength Training

INTERVENTIONS:
Other: Conservational Physical Therapy and Proprioceptive Strength Training — The proprioceptive training cycle consist of squats, single leg stand, slide steps , forward and backward step, toe walking , heel walking , side sway etc.
  Arms: Proprioceptive Strength Training
Other: Conservational Physical Therapy and Core Instability Strength Training — Core stability is essential part of lower limb rehabilitation; it is also known protocol which includes group of exercises in both standing and sitting improving biomechanics and functional performance of the body.
  Arms: Core Instability Strength Training

SUMMARY:
This study aims to determine the influence of core instability exercises in comparison to proprioceptive training in relieving pain, improving balance and physical function in general population of knee Osteoarthritis. The objective is to achieve beneficial results of interventions which can be used in betterment of treatment plan.

DETAILED DESCRIPTION:
A randomized control trial will be held at Safi hospital Faisalabad after the approval of the synopsis. The study will be double blinded clinical trial. Simple lottery method will be practiced to allocate subjects into two groups. Subjects are selected according to there explained inclusion exclusion criteria. The two groups are differentiated as control group and experimental group. Both the groups will be given the baseline intervention including TENS and Infrared. Along with baseline treatment control group will be given proprioceptive training and experimental group will be given core instability exercises. The evaluation is done before the research begin, after 6 weeks, after 12th week and Follow up on 16th week at the end of therapy. The outcomes will be assessed through Visual Analog Scale, Western Ontario and McMaster Universities Arthritis Index and Fullerton Advanced Balance scale. The data will be recorded pre and post treatment and compared after 12th week. Informed consent should be signed by each patient and analysis is done by Statistical Package of Social Sciences Version 21.

ELIGIBILITY:
Inclusion Criteria:

* Knee Osteoarthritis disease
* Kellgren Lawrence stage 1 to stage 4
* Unilateral or Bilateral Knee Osteoarthritis
* Patient who are willing to participate

Exclusion Criteria:

* History of any neurological condition e.g. Parkinson or vertigo.
* History of any past surgical procedure related to lower extremity.
* History of any chronic disease (hepatic, cardiac or renal diseases) which can affect the exercise training.
* History of severe orthopedic issues like fractures which may interfere in treatment sessions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Kellgren Lawrence scale | 12th Week
  Kellgren-Lawrence classification is typically applied within the context of knee Osteoarthritis. Based on the radiographic features, the severity of Osteoarthritis is given a grade from 0 to 4, with grade 0 signifying no presence of Osteoarthritis and grade 4 signifying severe Osteoarthritis.
Visual Analogue Scale | 12th Week
  Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
Fullerton Advanced Balance Scale | 12th Week
  The Fullerton Advanced Balance Scale assesses both static and dynamic balance under varying sensory conditions. Balance is measured in this test in active older adults who have higher levels of function.
Western Ontario and Mc Master Universities osteoarthritis Scale | 12th Week
  The Western Ontario and McMaster Universities osteoarthritis scale is widely used to assess pain, stiffness, and function in patients with osteoarthritis of the hip or knee.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No